CLINICAL TRIAL: NCT05767996
Title: School-based Education and Screening Program With Lipid Screening as a Means to Identify Familial Hyperlipidemia
Status: Enrolling by invitation | Type: Observational
Sponsor: Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Gary J. Luckasen, MD, Principal Investigator, University of Colorado Health
Other Study IDs: 20-6010
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Familial Hyperlipidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determination of FH status by genetic testing in school age children who have demonstrated elevated cholesterol on baseline screening.

ELIGIBILITY:
Inclusion Criteria:

Elevated cholesterol on baseline screening to use as means of identifying those with an FH variant

Exclusion Criteria:

* normal cholesterol

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Elementary school children participating in baseline biometric screening, including cholesterol; with those with elevated cholesterol receiving genetic testing to identify presence/absence of FH variant
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
School-based Education and Screening Program With Lipid Screening as a Means to Identify Familial Hyperlipidemia | Evaluation of family members over a defined 5 year period
  Percentage of school children who have elevated cholesterol related to FH variant

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States